CLINICAL TRIAL: NCT00343213
Title: Diagnostic and Prognostic Value of p16INK4a Expression in Low Grade Squamous Intraepithelial Lesions of the Cervix. Immunohistochemical Study on Biopsies (Retrospective and Prospective Analysis) and on Liquid Based (SurePath) Cervical Cytology (Prospective Analysis). Correlation With HPV Typing and Clinical Outcome.
Brief Title: Diagnostic and Prognostic Value of p16INK4a Expression in Low Grade Squamous Intraepithelial Lesions of the Cervix.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Christine GEILLER, Directeur de la Recherche Clinique et des Innovations, Hôpitaux Universitaires de Strasbourg
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 3454
Record Dates: First submitted 2006-06-21; First posted 2006-06-22 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 1 (CIN 1)
Keywords: Prognostic value of p16INK4a; CIN 1; LSIL; HPV
MeSH Terms: interventions — Colposcopy

INTERVENTIONS:
Procedure: colposcopy

SUMMARY:
P16INK4a has recently been described as a surrogate marker for HR-HPV associated squamous and glandular intraepithelial lesions of the cervix. The immunohistochemical staining pattern of p16INK4a in high grade intraepithelial neoplasia of the cervix (CIN 2 and 3) is diffuse, whereas in CIN 1 different staining patterns (diffuse, sporadic, focal or negative) can be seen. The aim of our study is to find out whether the p16INK4a staining pattern of CIN 1 is able to predict the outcome of the lesion. The retrospective part of the study includes cervical biopsies of 200 patients with CIN 1 and clinical follow-up for at least 5 years. p16INK4a staining and HPV detection by IHC will be correlated to clinical outcome.The prospective part of the study includes 300 patients with CIN 1 and LSIL on cytology. HPV detection by HCII and p16INK4a immunohistochemistry on liquid based cytology samples as well as p16INK4a staining and HPV detection by ISH on colposcopy guided biopsies will be correlated to clinical follow-up and colposcopy findings. Slides are analysed by 2 pathologists without knowledge of clinical data.

ELIGIBILITY:
Responsible women > 18 years with histologically proven CIN 1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-06

PRIMARY OUTCOMES:
p16INK4a staining pattern and HPV status of the initial biopsy

SECONDARY OUTCOMES:
p16INK4a staining pattern and histologic diagnosis of follow-up biopsies correlated with colposcopic findings.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Baldauf, MD, Study Director — Département de Gynécologie-Obstétrique - Hôpital de Hautepierre - Strasbourg - France
Locations (3):
- France (3):
  - Service de Gynécologie-Obstétrique - Centre Hospitalier Général, Haguenau
  - Service de gynécologie-obtétrique - Centre Hospitalier Général, Saverne
  - Département de Gynécologie-Obstétrique - Hôpital de Hautepierre, Strasbourg